CLINICAL TRIAL: NCT02893072
Title: Individualized Medical Nutrition Therapy Intervention Program for Women With Gestational Diabetes
Brief Title: Medical Nutrition Therapy Intervention Program for Women With Gestational Diabetes--a Prospective Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YYK-2016-002
Record Dates: First submitted 2016-08-23; First posted 2016-09-08 (Estimated); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Diabetes, Gestational
Keywords: Diabetes, Gestational; Nutrition Therapy
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Individualized medical nutrition therapy (Experimental): A comparison of normal lifestyle and medical nutrition therapy after intervention in the same individual
  Interventions: Behavioral: Individualized medical nutrition therapy

INTERVENTIONS:
Behavioral: Individualized medical nutrition therapy — The intervention group involves dietary and exercise advice and monitoring.

SUMMARY:
Gestational diabetes mellitus (GDM) is one of the most frequent complications of pregnancy, that affect between 1 to 14% of population around the world. The overall purpose of this study is to determine the efficacy of individualized medical nutrition therapy (MNT) intervention to reduce and control the development of GDM.

DETAILED DESCRIPTION:
The number of women with gestational diabetes mellitus had been increasing. Maternal GDM has a great impact on both the health of the mothers and the offspring. Antenatal lifestyle interventions, in particular dietary intervention appear to be feasible to improve maternal GDM and weight gain. To the best of our knowledge, there has been no such trial examining the feasibility of MNT intervention in pregnant women in Hu'nan province. The aim of this study is to evaluate the efficacy of individualized MNT intervention to reduce and control the development of GDM. This is a prospective study, 500 patients who meet inclusion and exclusion criteria will be included. The changes of glucose and weight will be evaluated every two weeks.

ELIGIBILITY:
Inclusion Criteria:

* Women with gestational diabetes

Exclusion Criteria:

* None

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 600 (Estimated)
Dates: Start 2015-11; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
intravenous glucose | every two weeks, from date of randomization until the date of parturition, assessed up to 10 months
  Investigators will measure the participants' intravenous glucose every two weeks.From date of randomization until the date of parturition,assessed up to 10 months.

CONTACTS AND LOCATIONS:
Overall Officials: Min Liu, M.D., Study Director — specify unaffiliated
Locations (1):
- the Third Xiangya Hospital of Central South University, Changsha, Hu'nan, China

IPD SHARING:
Plan to Share IPD: Yes
During and after our experiment, investigators will share the development in the website.
Supporting Information: Study Protocol
Time Frame: The data will be available in June 2018.
Access Criteria: Every body can get the information we shared.